CLINICAL TRIAL: NCT01701284
Title: A Randomized Open-Label Pilot Trial To Evaluate The Safety And Efficacy Of Repetitive Transcranial Magnetic Stimulation In Cancer Patients With Depression And Anxiety
Brief Title: Repetitive Transcranial Magnetic Stimulation in Cancer Patients With Depression and Anxiety
Acronym: rTMSinCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Neuronetics (Other)
Responsible Party: Principal Investigator, Mehmet Dokucu, Assistant Professor of Psychiatry, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 12CC12; NCI-2012-01691 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cancer in Remission (Any Type or Stage); Depression; Anxiety
Keywords: repetitive Transcranial Magnetic Stimulation; Cancer Survivors; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Transcranial Magnetic Stimulation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right-Sided Low-Frequency rTMS (Experimental): Participants will have rTMS administered at 1Hz to the right dorsolateral Prefrontal Cortex (dlPFC) once a day for 40 minutes, 5 days a week, for a total of six weeks.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Left-Sided High-Frequency rTMS (Experimental): Participants will have rTMS administered at 10Hz to the left dorsolateral Prefrontal Cortex (dlPFC) once a day for 40 minutes, 5 days a week, for a total of six weeks.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
  Other Names: Neurostar TMS Therapy(R) System

SUMMARY:
Cancer is a leading cause of mortality and morbidity worldwide. In addition, cancer is associated with high rates of depression and anxiety among its sufferers, and cancer patients with depression usually have worse treatment outcomes and long-term survival. Surprisingly, many cancer patients with depression do not receive treatment for their depression, perhaps because treatments for cancer-related depression are usually adapted from those used in non-cancer populations and may not be suitable for cancer patients. Moreover, cancer patients with depression are more likely to have a long latency of anti-depressant drug action, negative drug-drug interactions with cancer chemotherapies and an increased susceptibility for systemic side effects. Repetitive transcranial magnetic stimulation (rTMS) is a new treatment modality for depression that affects the brain directly with no systemic side effects and poses no potential for drug-drug interactions. rTMS therapy was recently cleared by the FDA as an antidepressant treatment for treatment-resistant Major Depressive Disorder, and now is being evaluated for a wide array of additional psychiatric indications. This randomized, open label, two-arm, pilot study will investigate the safety, tolerability, feasibility and the efficacy of two forms of rTMS (i.e., left (fast) and right (slow) sided rTMS) in cancer-related depression. The study hypotheses are that rTMS will significantly reduce symptoms of depression and that right-sided slow rTMS will be more effective than left-sided fast rTMS for the treatment of severe anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 22-80
* Had a previous diagnosis of cancer (any type or stage) confirmed by official medical records
* Has a DSM IV diagnosis of Major Depressive Disorder
* Has a HAM-D 24-item score of more than 20
* Failed to receive satisfactory improvement from one prior antidepressant medication at or above the minimal effective dose and duration in the current depressive episode
* All participants must have given signed, informed consent prior to registration in study

Exclusion Criteria:

* Participant had breast cancer with brain metastases
* There is evidence of the disease at the time of entry into the trial
* Presence or recent history of other concurrent cancers, with the following exceptions:

  * Participants with completely treated basal or squamous skin cancers can be included in the study if their physicians deem that they are medically stable
  * Participants with completely treated in situ carcinoma of the breast or cervix may be included in the study if they have not had chemotherapy within the past month and their physicians deem that they are medically stable
  * Participants with pre-cancerous lesions in the colon can be included in the study if they have not had chemotherapy within the past month and their physicians deem that they are medically stable
* Participant had recent surgery (within two weeks)
* Participant is undergoing chemotherapy
* Participant is pregnant or nursing
* Participant has any metallic object in or around their head
* Participant has a pacemaker
* Has unstable suicidal ideation as determined by the patient's treating psychiatrist
* Substance use disorder within the prior six months
* Significant history of head injury/trauma as defined by loss of consciousness for more than 1 hour
* Recurring seizures resulting from the head injury
* Clear cognitive sequelae from the head injury and cognitive rehabilitation following the injury
* Any disorder that would predispose the participant to seizures
* Use of concomitant medications that substantially increase seizure risk. Such drugs could include neuroleptics (ex. haloperidol, droperidol), clozapine, tricyclic antidepressants (ex. amoxapine, clomipramine), bupropion (particularly the immediate release - IR - formulation) donepezil, psychostimulants (ex. methylphenidate), theophylline and/or other drugs that reduce the seizure threshold. For individuals on any of these medicines, a study clinician will evaluate the drugs and doses to determine the risks and benefits. These will then be discussed with the individual's Primary Care Physician to determine if the individual should be excluded from the study.

Ages: 22 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Overall change in depression severity | 0, 2, 4, and 6 weeks
  Overall change in depression severity (as measured by the Hamilton Depression Rating Scale) will be measured for each treatment arm.
Relative change in depression severity | 0, 2, 4, and 6 weeks
  Change in depression severity (as measured by the Hamilton Depression Rating Scale) for a treatment arm will be compared relative to change in depression severity in the other treatment arm.
Presence and changes in severity of side effects | 0, 2, 4, and 6 weeks
  At weeks 2, 4 and 6, UKU Side Effects Rating Scale scores will be compared to baseline UKU scores to determine changes in presence and severity of side effects. Additionally, UKU scores at weeks 2, 4, and 6 will be used to determine probability that side effects are related to intervention.

SECONDARY OUTCOMES:
Overall change in anxiety severity | Weekly (starting with week 0 through week 6)
  Overall change in anxiety severity (as measured by the Hamilton Anxiety Rating Scale) will be measured for each treatment arm.
Relative change in anxiety severity | Weekly (starting with week 0 through week 6)
  Change in anxiety severity (as measured by the Hamilton Anxiety Rating Scale) for a treatment arm will be compared relative to change in anxiety severity in the other treatment arm.
Correlation of anxiety with change in depression severity | 0 and 6 weeks
  Baseline anxiety severity (as measured by the Hamilton Anxiety Rating Scale) will be correlated with change (from baseline to end of week 6) in depression severity (as measured by the Hamilton Depression Rating Scale) for each treatment arm and compared.
Correlation of anxiety with harm avoidance personality trait | Baseline
  Baseline anxiety severity (as measured by the Hamilton Anxiety Rating Scale) will be correlated with Harm Avoidance scores from the TCI personality inventory

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Dokucu, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgess C, Cornelius V, Love S, Graham J, Richards M, Ramirez A. Depression and anxiety in women with early breast cancer: five year observational cohort study. BMJ. 2005 Mar 26;330(7493):702. doi: 10.1136/bmj.38343.670868.D3. Epub 2005 Feb 4. PMID 15695497
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] Janicak PG, O'Reardon JP, Sampson SM, Husain MM, Lisanby SH, Rado JT, Heart KL, Demitrack MA. Transcranial magnetic stimulation in the treatment of major depressive disorder: a comprehensive summary of safety experience from acute exposure, extended exposure, and during reintroduction treatment. J Clin Psychiatry. 2008 Feb;69(2):222-32. doi: 10.4088/jcp.v69n0208. PMID 18232722
- [Background] Machado S, Paes F, Velasques B, Teixeira S, Piedade R, Ribeiro P, Nardi AE, Arias-Carrion O. Is rTMS an effective therapeutic strategy that can be used to treat anxiety disorders? Neuropharmacology. 2012 Jan;62(1):125-34. doi: 10.1016/j.neuropharm.2011.07.024. Epub 2011 Jul 27. PMID 21807002
- [Background] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044
- [Background] Paes F, Machado S, Arias-Carrion O, Velasques B, Teixeira S, Budde H, Cagy M, Piedade R, Ribeiro P, Huston JP, Sack AT, Nardi AE. The value of repetitive transcranial magnetic stimulation (rTMS) for the treatment of anxiety disorders: an integrative review. CNS Neurol Disord Drug Targets. 2011 Aug;10(5):610-20. doi: 10.2174/187152711796234943. PMID 21631403
- [Background] Schutter DJ. Antidepressant efficacy of high-frequency transcranial magnetic stimulation over the left dorsolateral prefrontal cortex in double-blind sham-controlled designs: a meta-analysis. Psychol Med. 2009 Jan;39(1):65-75. doi: 10.1017/S0033291708003462. Epub 2008 Apr 30. PMID 18447962
- [Background] Slotema CW, Blom JD, Hoek HW, Sommer IE. Should we expand the toolbox of psychiatric treatment methods to include Repetitive Transcranial Magnetic Stimulation (rTMS)? A meta-analysis of the efficacy of rTMS in psychiatric disorders. J Clin Psychiatry. 2010 Jul;71(7):873-84. doi: 10.4088/JCP.08m04872gre. Epub 2010 Mar 9. PMID 20361902